CLINICAL TRIAL: NCT04669041
Title: A Randomized Double-blinded, Double Dummy, Active-controlled, Parallel Design, Phase 3 Clinical Trial to Evaluate the Efficacy and the Safety of Single Pill Combination (SPC) Ezetimibe/Rosuvastatin in Chinese Adult Patients With Primary Hypercholesterolemia, Not Adequately Controlled on Statin Therapy
Brief Title: A Study to Evaluate the Efficacy and the Safety of Single Pill Combination (SPC) Ezetimibe/Rosuvastatin in Chinese Adult Patients With Primary Hypercholesterolemia Not Adequately Controlled on Statin Therapy
Acronym: ROZEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPS16135; U1111-1227-3920 (Other: UTN)
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single pill combination (SPC) (Experimental): Once daily rosuvastatin 10 mg for 4 weeks, then once daily SPC ezetimibe 10 mg /rosuvastatin 10 mg (E10/R10) for 8 weeks
  Interventions: Drug: Rosuvastatin; Drug: SPC ezetimibe/rosuvastatin; Drug: Placebo
- Rosuvastatin (Active Comparator): Once daily rosuvastatin 10 mg for 4 weeks, then once daily rosuvastatin 10 mg (R10) for 8 weeks
  Interventions: Drug: Rosuvastatin; Drug: Rosuvastatin active capsule; Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Pharmaceutical form:Tablet Route of administration: Oral
  Other Names: Crestor®
Drug: SPC ezetimibe/rosuvastatin — Pharmaceutical form:Tablet Route of administration: Oral
  Arms: Single pill combination (SPC)
Drug: Rosuvastatin active capsule — Pharmaceutical form:Capsule Route of administration: Oral
  Arms: Rosuvastatin
Drug: Placebo — Pharmaceutical form:Tablet Route of administration: Oral
  Arms: Rosuvastatin
Drug: Placebo — Pharmaceutical form:Capsule Route of administration: Oral
  Arms: Single pill combination (SPC)

SUMMARY:
Primary Objective:

To demonstrate the superiority of the single pill combination (SPC) ezetimibe 10 mg/rosuvastatin 10 mg (E10/R10) compared to rosuvastatin 10 mg (R10), in the reduction of low density lipoprotein cholesterol (LDL-C) after 8 weeks.

Secondary Objectives:

* To evaluate the proportion of patients who attain their LDL-C goal.
* To evaluate the effect of SPC (E10/R10) compared to rosuvastatin 10 mg (R10) in reduction of LDL-C at Week 4.
* To evaluate the effect of SPC (E10/R10) compared to R10 on other lipid parameters at Week 4 and Week 8.
* To evaluate the safety of SPC (E10/R10) and R10.

DETAILED DESCRIPTION:
Study duration per participants is approximatively 16 weeks.

ELIGIBILITY:
Inclusion criteria :

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Patients with primary hypercholesterolemia.
* Inclusion criteria in the run-in period: Participants who are not adequately controlled (defined by screening LDL-C >2.6 mmol/L (100 mg/dL) and ≤4.9 mmol/L (190 mg/dL)with a 10 mg stable daily dose of rosuvastatin, or equipotent statin for 4 weeks prior to the screening visit, without any other lipid modifying therapy (LMT). Inclusion criteria in the randomized double-blind period: Participants who are not adequately controlled based on sample taken at qualifying pre randomization visit, despite stabilized dose of rosuvastatin 10 mg (defined by measured LDL-C ≥2.6 mmol/L (100 mg/dL) and ≤4.9 mmol/L (190 mg/dL).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion criteria:

* Homozygous familial hypercholesterolemia (FH) (clinically or previous genotyping).
* Patient who has received LDL-C plasmapheresis treatment within 2 months prior to the screening visit, or has plans to receive it during the study.
* Recently diagnosed (within 3 months prior to the screening visit) myocardial infarction (MI), unstable angina, myocardial revascularization (percutaneous coronary intervention [PCI], coronary artery bypass graft surgery [CABG]), transient ischemic attack (TIA), or stroke, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease.
* Planned to undergo scheduled PCI, CABG, carotid or peripheral revascularization during the study.
* Severe hypertension (treated or untreated) with systolic blood pressure (SBP) >160 mm Hg or diastolic blood pressure (DBP) >100 mm Hg at study entry.
* History of severe congestive heart failure (New York Heart Association Class IIIb or IV) within the past 12 months.
* Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins, according to Investigator's medical judgement.
* Uncontrolled (as determined by fasting glucose >180 mg/mL or HbA1c >9%) or newly diagnosed (within 3 months of study entry) diabetes mellitus at the screening visit.
* History of cancer within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* Conditions/situations such as:

  * Patient with a short life expectancy.
  * Patient with conditions/concomitant diseases making them non-evaluable for the primary efficacy endpoint, according to Investigator's medical judgement.
  * Requirement for concomitant treatment that could bias primary evaluation, according to Investigator's medical judgement.
  * Impossibility to meet specific protocol requirements (eg, ability to make study visits).
  * Patient is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the study.
  * Patient not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.
* Known history of hypersensitivity reaction to statins and/or ezetimibe.
* Current myopathy.
* A history of statin-induced myopathy or rhabdomyolysis.
* Current active liver disease including unexplained, persistent elevations of serum transaminases and any serum transaminase elevation exceeding 3 x upper limit of normal (ULN) range at the screening visit.
* All contraindications to the active comparator (rosuvastatin) and background therapies or warning/precaution of use (when appropriate) as displayed in the respective National Product Labeling.
* Patients not previously instructed on a cholesterol-lowering diet prior to the screening visit.
* Use of systemic corticosteroids, unless used as replacement therapy for pituitary/adrenal disease with a stable regimen for at least 6 weeks prior to screening visit.
* Use of hormone replacement therapy or oral contraceptives unless regimen has been stable in the past 6 weeks prior to the screening visit and no plans to change the regimen during the study.
* Concomitant administration of cyclosporine (at screening and randomization visits).
* Human immunodeficiency virus (HIV) patients receiving protease inhibitors (at screening and randomization visits).
* Patient who has taken any active investigational drugs (E10/R10) within 1 month or 5 half-lives prior to screening, whichever is longer.
* Laboratory findings obtained during the screening visit (V1):

  * Fasting serum TGs >400 mg/dL.
  * Positive serum pregnancy test.
  * Serum creatine kinase >3 times ULN.
  * Thyroid-stimulating hormone (TSH) < lower limit of normal (LLN) or > ULN.
  * Glycated hemoglobin A1c (HbA1c) >9%.
  * Estimated glomerular filtration rate <30 mL/min/1.73 m2.
  * Alanine aminotransferase or AST >3 x ULN.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or subjects who are legally institutionalized.
* Any technical/administrative reason (eg, patient homeless) that makes it impossible to enroll/randomize the patient in the study.
* Alcohol abuse according to Investigator's medical judgement.
* Participants are dependent on the Sponsor or Investigator (in conjunction with Section 1.61 of the ICH-GCP Ordinance E6).
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.
* Any specific situation during study implementation/course that may rise ethics considerations.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Percent change in measured LDL-C from baseline (the last available measured LDL-C value obtained up to randomization) to Week 8 | Baseline to Week 8
  The percent change from baseline in measured LDL-C at Week 8 will be analyzed in the modified intent-to-treat (mITT) population using a mixed effect model with repeated measures (MMRM) approach.

SECONDARY OUTCOMES:
Proportion of patients who attain lipid goal (measured LDL-C <2.6 mmol/L [100 mg/dL]) at Week 8 | Week 8
Percent change in measured LDL-C plasma level from baseline to Week 4 | Baseline to Week 4
Percent change in total cholesterol (TC) from baseline to Week 8 | Baseline to Week 8
Percent change in TC from baseline to Week 4 | Baseline to Week 4
Percent change in triglyceride (TG) serum levels from baseline to Week 8 | Baseline to Week 8
Percent change in TG serum levels from baseline to Week 4 | Baseline to Week 4
Percent change in high density lipoprotein cholesterol (HDL-C) from baseline to Week 8 | Baseline to Week 8
Percent change in HDL-C from baseline to Week 4 | Baseline to Week 4
Number of patients with adverse events (AEs) | Up to 16 weeks (±3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- China (40):
  - Investigational Site Number :1560033, Baotou
  - Investigational Site Number :1560001, Beijing
  - Investigational Site Number :1560068, Beijing
  - Investigational Site Number :1560021, Beijing
  - Investigational Site Number :1560025, Bengbu
  - Investigational Site Number :1560045, Changchun
  - Investigational Site Number :1560067, Changchun
  - Investigational Site Number :1560052, Changsha
  - Investigational Site Number :1560041, Chengdu
  - Investigational Site Number :1560060, Chongqing
  - Investigational Site Number :1560015, Dalian
  - Investigational Site Number :1560029, Haikou
  - Investigational Site Number :1560006, Hohhot
  - Investigational Site Number :1560007, Hohhot
  - Investigational Site Number :1560014, Jilin
  - Investigational Site Number :1560020, Jinan
  - Investigational Site Number :1560061, Lishui
  - Investigational Site Number :1560071, Liuchow
  - Investigational Site Number :1560066, Nanjing
  - Investigational Site Number :1560055, Nanning
  - Investigational Site Number :1560027, Shanghai
  - Investigational Site Number :1560034, Shenyang
  - Investigational Site Number :1560010, Siping
  - Investigational Site Number :1560002, Tianjin
  - Investigational Site Number :1560053, Tianjin
  - Investigational Site Number :1560047, Wuhan
  - Investigational Site Number :1560009, Wuhan
  - Investigational Site Number :1560035, Wuhan
  - Investigational Site Number :1560022, Xi'an
  - Investigational Site Number :1560070, Xi'an
  - Investigational Site Number :1560003, Xuzhou
  - Investigational Site Number :1560065, Yangzhou
  - Investigational Site Number :1560057, Yanji
  - Investigational Site Number :1560064, Yinchuan
  - Investigational Site Number :1560019, Yueyang
  - Investigational Site Number :1560062, Yuncheng
  - Investigational Site Number :1560005, Zhanjiang
  - Investigational Site Number :1560011, Zhenjiang
  - Investigational Site Number :1560063, Zhuzhou
  - Investigational Site Number :1560037, Zibo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Su Q, Liu Y, Zhang G, Xu L, Wang M, Mei S, Garon G, Wu Y, Lv Q, Ma C. Efficacy and Safety of Single-Pill Combination of Rosuvastatin and Ezetimibe in Chinese Patients with Primary Hypercholesterolemia Inadequately Controlled by Statin Treatment (ROZEL): A Randomized, Double-Blind, Double Dummy, Active-Controlled Phase 3 Clinical Trial. Adv Ther. 2023 Dec;40(12):5285-5299. doi: 10.1007/s12325-023-02666-z. Epub 2023 Sep 28. PMID 37770770
- See also: LPS16135 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25279&tenant=MT_SNY_9011